CLINICAL TRIAL: NCT00495716
Title: Effect of Suppressive Therapy on Behavioral Determinants of HSV-2 Transmission
Brief Title: Effect of HSV-2 Suppressive Therapy on Sexual Behavior
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator relocated and study funding ended.
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Anna Wald, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 32545; K23AI071257-01A1 (NIH)
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Episodic Treatment Arm (Active Comparator): 800 mg acyclovir orally 3 times daily for 2 days at the start of a genital herpes recurrence
  Interventions: Drug: acyclovir
- Suppressive Therapy Arm (Active Comparator): 400 mg acyclovir orally twice daily for 1 year
  Interventions: Drug: acyclovir

INTERVENTIONS:
Drug: acyclovir — 800 mg acyclovir orally 3 times daily for 2 days at the start of a genital herpes recurrence
  Arms: Episodic Treatment Arm
Drug: acyclovir — 400 mg acyclovir orally twice daily for 1 year
  Arms: Suppressive Therapy Arm

SUMMARY:
The purpose of this study is to determine what effect suppressive therapy has on sexual behavior and quality of life among persons with genital herpes (HSV) who have multiple sex partners.

Study terminated; investigator relocated and study funding ended. Results were never analyzed because data were not collected.

DETAILED DESCRIPTION:
We plan to conduct a randomized controlled trial of chronic suppressive acyclovir, 400 mg orally twice daily (standard dose) versus episodic acyclovir for treatment of genital herpes recurrences. We will enroll 500 HSV-2 seropositive single persons (250 per arm), stratified by gender and history of symptomatic genital herpes, and prospectively follow them for 1 year to assess sexual behavior, adherence to therapy, and herpes-related quality of life. These outcomes will be measured by self-report in a confidential, computer-based assessment. We plan to use data from this trial to model the effect that increasing the proportion of sexually-active HSV-2 infected persons taking suppressive therapy will have on population-level incidence and prevalence of HSV-2.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* HSV-2 seropositive by Western blot OR documented culture positive for HSV-2 from anogenital site
* 2 or more vaginal or anal sex partners in the past 12 months
* Not currently in a monogamous sexual relationship of >= 6 months duration
* Willing and able to be randomized and comply with the study protocol

Exclusion Criteria:

* Pregnancy or intention to become pregnant within the next year
* Suppressive therapy with acyclovir, valacyclovir, or famciclovir within 2 weeks of enrollment/randomization
* 6 or more symptomatic herpes recurrences in the prior 12 months or in the 12 months prior to starting suppressive therapy if on suppressive therapy during the prior 12 months
* HIV seropositive or known immunocompromising medical condition. HIV negative test must be performed within 60 days of Visit 1 (enrollment/randomization). For current or former participants in HIV vaccine clinical trials for whom HIV vaccine-induced seropositivity potentially leading to vaccine study unblinding may be a concern, a report from the Seattle HVTU documenting that the participant is HIV uninfected based on HIV testing done within 60 days of Visit 1 will be accepted in lieu of HIV testing done at our clinic.
* Intention to move from the Seattle area within the next year
* Known allergy, intolerance, or medical contraindication to acyclovir
* Inability to understand, speak, and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wald, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Episodic Treatment Arm | Suppressive Therapy Arm
Started | 35 | 37
Completed | 20 | 24
Not Completed | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Episodic Treatment Arm | Suppressive Therapy Arm | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Continuous [Mean (Full Range); unit: years] | 40 [18 to 79] | 39 [22 to 63] | 39 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 21 | 22 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 12 | 24
  White | 21 | 25 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Suppressive Antiviral Therapy on Sexual Behavior Among HSV-2 Seropositive Persons With Multiple Sexual Partners.
Time Frame: 1 year
Population: Study terminated; investigator relocated and study funding ended. Results cannot be analyzed because data were not collected.
Arm/Group | Episodic Treatment Arm | Suppressive Therapy Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Episodic Treatment Arm | Suppressive Therapy Arm
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37
Other Adverse Events (participants affected / at risk) | 0/35 | 0/37

LIMITATIONS AND CAVEATS:
Study terminated; investigator relocated and study funding ended. Results cannot be analyzed because data were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes